# University of Minnesota

# **HEALTH & BIOLOGICAL/MEDICAL APPLICATION FORM**

Version 6.2

Updated January 2015, check <a href="http://www.irb.umn.edu">http://www.irb.umn.edu</a> for the latest version

Route this form to:

U Wide Form: UM 1571

See instructions below.

Jan. 2015

| Submit this application, along with all required appendices and supplemental documents to the University of Minnesota IRB | | | IRB Use Only IRB Study # Click here to enter text. |
|---|---|---|---|
| PI must submit request using MMC 820 University of Minnesota e-mail 420 Delaware St. SE Account. Academic advisor and/or Co- | Human Research Protection Program MMC 820 420 Delaware St. SE | | For more information please visit our website http://www.research.umn.edu/irb/index.html Contact our office Phone: 612-626-5654 Email: irb@umn.edu Fax: 612-626-6061 |
| Project Title | | | |
| If the project is funded, the Sponsored Project Admi<br>the project is funded by multiple grants, provide all | • | | oject title must match the IRB project title. If |
| Transversus Abdominis Plane (TAP) Infiltration vs. Surgical Infiltration of Local Anesthetic in Laparoscopic and Robotic assisted Hysterectomy | | | |
| Section 1 Principal Investigator | | | |
| Name | | Highest | Earned Degree: |
| Geller, Melissa A | | MD | |
| Preferred contact information: gelle005@umn.edu | | | |
| Preferred email or phone number at which the PI may be conta | icted by IRB st | aff or rev | iewers to resolve questions or concerns. |
| Affiliation and contact information | | | |
| ☑University of Minnesota (complete contact info section 1 on | ly) | | |
| Fairview (complete contact info section 2 only) | | | |
| Gillette (complete contact info section 2 only) | | | |
| Required Contact information U of M Internet ID (x.500): | gelle005 | | |
| Carrier 4 Haffa ada | | | |
| Section 1 - U of M only U of M Employee/student II Number: | | | |
| University Department: | University Department: Department | | ment of Obstetrics, Gynecology and Women's |
| | Health, Divisio | | of Gynecologic Oncology |
| Required contact information Address: | Address: | | one number: |
| Section 2 Non-U of M only | | | |
| | | | Mobile Pager Office |
| | | | ail address: |

| Occupational Position: | | |
|---|---|---|
| ☑Faculty ☐Physician ☐Staff ☐Student - Student | dents must complete the faculty academi | c advisor section below and submit Appendix J |
| Other: | | |
| Conflict of Interest: | | |
| Does the PI have a reportable conflict as defined | in Section 11 of the application? | |
| ☐Yes ⊠ No | | |
| Required CITI Human Subjects Training | | HIPAA TRAINING |
| Date (Month/Year) CITI completed (either initial of | or refresher course): | Check box below if HIPAA training is required. |
| | | ☐ HIPAA Required – Data contains PHI |
| Note: The IRB requires researchers to complete re completion of initial course. For more information | | HIPAA Training completed through: |
| Training | on training requirements see <u>mb</u> | ⊠ UMN |
| | | Other: |
| For information regarding human subjects of | and HIPAA training requirements ple | ase go to http://www.irb.umn.edu/training.html, |
| As Principal Investigator of this study, I assure the | e IRB that the following statements are | true: |
| The information provided in this form is | correct. | |
| I have evaluated this protocol and deter | rmined that I have the resources necessa | ry to protect participants, such as adequate |
| funding, appropriately trained staff, and | d necessary facilities and equipment. | |
| • I will seek and obtain prior written approval from the IRB for any substantive modifications in the proposal, including changes in procedures, co-investigators, funding agencies, etc. | | |
| <ul> <li>I will promptly report any unexpected or otherwise significant adverse events or unanticipated problems or incidents that may<br/>occur in the course of this study.</li> </ul> | | |
| <ul> <li>I will report in writing any significant new findings which develop during the course of this study which may affect the risks and<br/>benefits to participation.</li> </ul> | | |
| I will not begin my research until I have received written notification of final IRB approval. | | |
| I will comply with all IRB requests to report on the status of the study. | | |
| I will maintain records of this research according to IRB guidelines. | | |
| <ul> <li>The grant that I have submitted to my funding agency which is submitted with this IRB submission accurately and completely reflects what is contained in this application.</li> </ul> | | |
| If these conditions are not met, I understand that approval of this research could be suspended or terminated. | | |
| | MD | Today's date. |
| Signature/Digital signature/x.500 of PI | Title of PI | Date |
| Faculty Academic Advisor - Student Research If the PI of this research is a student, include Appendix J filled out by the advisor with this application form. | | |
| Student research requires the approval of a faculty academic advisor. As academic advisor to the student investigator, the advisor assumes responsibility for ensuring that the student complies with University policies and federal regulations regarding the use of human subjects in | | |

Faculty Academic Advisor Name (Last name, First name MI):

**University Department:** 

| U of M Employee ID: | U of M x.50 | 0 ID (ex. smith001): |
|---|---|---|
| Conflict of Interest: Does this person have a reportable conflict as defined in Section 11 of the application? Yes No | | |
| Human Subjects Training: | | HIPAA TRAINING |
| CITI – Date completed (either initial or refresher course): | | Check box below if HIPAA training is required. HIPAA Required – Data contains PHI |
| Note: The IRB requires researchers to complete refreshers courses every three years after completion of initial course. For more information on training requirements see <a href="IRB Training">IRB Training</a> | | HIPAA Training completed through: UMN Other: |
| | Today's dat | e. |
| Signature/Digital signature/x.500 of Advisor<br>Advisor must be cc'ed on emailed submission to the IRB | Date | |
| Person preparing this document | | |
| PI prepared this application – section 1 complete | | |
| The person named below prepared this application | | |
| Name: Prefer | Name: Preferred contact info: | |
| Role on study: Co-Investigator Study Coordinator (Research Staff) | | |
| The person preparing the document must be listed on the application as a co-investigator or in a role that allows him/her to receive correspondence related to the application. See section 13 of the application for more information | | |
| Additional study personnel? Complete section 13 of this application. | | |
| Section 2 Summary of Activities | | |
| The following questions must be answered in lay language or language understood by a person unfamiliar with your area of research. A research plan or protocol is required with this submission. In the responses below, area-specific jargon should be avoided or explicitly explained. Do not say "see protocol" or "protocol attached". Protocol templates are available on the IRB forms page. | | |
| Trotocor templates are available on the into forms page. | | |

### 2.1 What is your research question?

State hypothesis or primary objective, and provide a brief background on subject population, treatment procedures, and the rationale for conducting the study.

This study aims to test whether there is a difference in the analgesic effect between TAP blocks and surgical infiltration during the first 72 hours following laparoscopic and robotic total hysterectomies.

Laparoscopic and Robotic assisted hysterectomy is a surgical procedure that is a minimally invasive way in which to remove the uterus, which has less scarring and fewer complications. However, this procedure, much like its open-surgical counterpart, is often associated with significant post-operative pain. To augment this pain there are many

different analgesic techniques available to offset pain. Ultrasound-guided transversus abdominis plane (TAP) block is one such procedure involving the injection of a local anesthetic into the plane of the transversus abdominal muscle where the terminal branches of nerves lie. A similar, yet different analgesic approach is that of direct injection of local anesthetic into the incision by the surgeon during or just after surgical procedures. These two approaches have both been proven to decrease post-operative pain in patients for many procedures, but never compared to one another.

### Background and Significance

Even with the advancement of using laparoscopic and robotic technologies in total hysterectomies, patients still suffer from pain. This study hopes to use a randomized controlled double-blinded approach to investigate the different analgesic outcomes from surgical infiltration of analgesics to that of ultrasound-guided transversus abdominis plane (TAP) blocks in this procedure.

Other studies have looked at the enhanced analgesic efficacy of both TAP blocks in laparoscopic and robotic procedures, as well as that of direct infiltration of anesthetics into the incisions following surgery.1 Up to this point, however, these two practices have not been undertaken in a single double-blind study in which to compare the analgesic efficacies.

| 2.2 Who developed the research plan/protocol? | | |
|---|---|---|
| Principal Investigator | Business and Industry Sponsor | Other: |

### 2.3 Explain how the study design and methods will answer the research question.

This is a double blinded randomized study. All patients will receive one form of local anesthetic pain relief either from TAP or infiltration. Patients will be randomized to one of two study arms in a double-blinded, placebo controlled study. All patients will receive a TAP infiltration and all patients will receive infiltration into the incision. In one arm the TAP infiltration will contain 10 mL of 0.25 % bupivacaine with epinephrine injected followed by 20 mL of a 50:50 mixture of liposomal bupivacaine and normal saline. This will then be repeated on the contralateral side. In the same arm the surgeon infiltration into the incision will consist of 10 ml of normal saline per port site, 5 ml prior to incision and 5 ml prior to closure at each port site.

In the second arm the bilateral TAP infiltration will consist of 30 mL of normal saline per side. In the same arm the surgeon infiltration will consist of 10 mL of 0.25% bupivacaine per port site. The surgeon infiltration will consist of 5 ml of 0.25% bupivacaine prior to incision and 5 ml of 0.25% bupivacaine prior to closure at each port site.

A TAP infiltration is an injection of local anesthetic under the covering of the transversus abdominis muscle layer which provides effective post operative analgesia.2-5 This layer is found using an ultrasound, which is a beam of high frequency sound that allows one to visualize images in the body. Then using this ultrasound we can see our needle as it pierces the covering of the transversus abdominis muscle layer and watch as the local anesthetic is infiltrated into this plane. This is done on both sides of the abdomen to provide analgesia to the skin, muscle, and facial layers of the abdomen. This is currently standard of care at our institution and will be performed within one hour of surgical incision. The injection will consist of 10 mL of 0.25% bupivacaine with epinephrine followed by 20 mL of liposomal bupivacaine saline mixture or 10 ml of saline followed by 20 ml of saline and then repeated on the contralateral side.

Surgical Infiltration of the study solution will be performed both prior to incision and at the end of surgery just prior to closure of incisions. At each time, the surgeon will inject 5 mL of 0.25% bupivacaine into each of the port site

| incisio | ons. | |
|---|---|---|
| Investigational Drug Service (IDS) pharmacy will be charged with the blinding of medications vs. saline for these procedures. | | |
| 2.4 W | hat will the subjects be asked to do solely for th | e purpose of this research? |
| Subjects will be asked to be randomly assigned to receive either a TAP with liposomal bupivacaine or infiltration with bupivacaine. They will also be asked to answer questions at various time points related to their pain, answer a survery on their quality of recovery. They will also be asked to allow the research staff to access their medical chart to obtain information about their pain medication use, complications, demographics, and time of discharge. | | |
| 2.5 D | oes the study involve treatment? | |
| | No. | |
| | Yes. List any procedure that would be performed if research was not conducted (i.e. procedures performed for diagnostic or treatment purposes). | |
| | all procedures would be performed if research was not conducted as both the TAP and infiltration are standard of care. | |
| | dicate whether your research includes any of the bmitted with your application: | e following to determine which supplemental forms must |
| If the | research includes | Appendices and supplemental materials required |
| | Administration of approved or unapproved drugs, chemical or biological agents | Appendix E required with the application |
| | Administration of approved or unapproved devices | Appendix F required with the application |
| | Genetic testing (whether or not results are returned to subjects) | Appendix G required with the application |
| | Use of (collecting or having access to) Protected Health Information (PHI) | Appendix H required with the application |
| | Field Work | Appendix L required with the application |
| | Use of a deceptive technique | Appendix N required with the application A debriefing script is also required. |
| | Community based participatory research | Appendix Q required with the application |
| | Collection or storage of biological samples | Appendix T required with the application |

| | (including blood draws, marrow biopsy sampling, biopsy of other tissues) | |
|---|---|---|
| | Use of Magnetic Resonance devices housed at the Center for Magnetic Resonance Research (CMRR) | Documentation of CMRR Safety Committee approval required. CMRR users must submit the completed CMRR Device and Safety Review form to the CMRR prior to submission of their IRB application. A draft copy of the IRB application must be included for CMRR Safety Committee review. Documentation of approval by the CMRR Safety Committee will be provided to the researcher to include with the IRB application. |
| | Potential biohazards including recombinant and synthetic nucleic acid, human gene transfer, biologically-derived toxins or infectious agents | Institutional Biosafety Committee approval required prior to final approval. If an IBC application has been submitted for this research, provide the study number. |
| | Biologically-derived toxins (including truncated or mutated toxins) | Institutional Biosafety Committee approval required prior to final approval. If an IBC application has been submitted for this research, provide the study number. |
| | Infectious agents (bacteria, viruses, protozoans, fungi) | Institutional Biosafety Committee approval required prior to final approval. If an IBC application has been submitted for this research, provide the study number. |
| | Use of radiation (x-ray imaging, radiopharmaceuticals, external beam or brachytherapy) | All University Radiation Protection Committee (AURPAC) approval required prior to final IRB approval. |
| Secti | on 3 Risks and Benefits | |
| 21 0 | ages indicate if the prepared research will in the | do any of the following (shock all that apply). The list |
| below | • • | de any of the following (check all that apply). The list ents or procedures in research with associated risks that |
| | Administration of physical stimuli | |
| | Probing for personal or sensitive information in surveys or interviews | |
| | Collection of data with identifiers | |

| | Possible invasion of privacy of the subject or the subject's family |
|---|---|
| | Modification or extension of a surgical process to achieve research related objectives. |
| | Major changes in diet, exercise, or sleep |
| | Manipulation of psychological or social variables such as sensory deprivation, social isolation, psychological stresses |
| | Placebo Use |
| | Treatment will be withheld or subjects will discontinue current treatment (a wash out period is included) |
| | None of the above |
| | scribe in detail the nature and degree of the risk associated with participation. The risks must be disclosed consent form. Include in the response all potential risks, not just those indicated in the checklist above. |
| placeb<br>saline. | is the potential of loss of privacy as the medical chart is accessed by the research staff. In addition there is a to used however no patient will be without pain medication. The TAP will either consist of local anesthetic or When the TAP consists of saline the infiltration will consist of local anesthetic and when the TAP consists of nesthetic the infiltration will consist of saline. |
| injecte | njection of local anesthetic there is risk of the block or infiltration not working. There is risk of it being ed in the wrong area and there is risk of local anesthetic toxicity albeit the dosages used are well below those would place the patient at risk of local anesthetic toxicity. |
| 3.3 De | scribe the precautions that will be taken to minimize each of the risks identified in questions 3.1 and 3.2. |
| | ient charts will be accessed by a trained research personnel. They will not record any identifiers. Patient's asked if they are willing to answer questions prior to each round of questions regarding pain scores and vs. |
| infiltra | P and infiltration are standard of care. Either or would be used if we were not doing the research. The TAP ation is performed by trained anesthesiologists and are under ultrasound real time guidance. The infiltration ormed by trained surgeons. |
| the sp | t any anticipated direct and societal benefits to participation in this research project. If none, state that in ace provided below and in the consent form. The benefit of receiving treatment is not necessarily a benefit ticipation in the research project. Compensation paid to subjects is not considered a benefit. |
| none | |
| 3.5 Jus<br>subjec | stify the risk in terms of the potential scientific yield and in relation to the anticipated benefits to the sts. |
| decrea | enefits of this study would be to find the most effective method of pain control which would not only ase patient's pain but decrease their use of opioids. As opioids are a significant burden on society in terms of e, addiction, and even death. It is important we find ways to minimize postoperative pain and postoperative |

| Secti | ion 4 Su | bject Profile | | | |
|---|---|---|---|---|---|
| sets n<br>appro | ecessary? wed by the | Subjects who go thr<br>IRB even if they hav | ough the consent<br>ve no further partic | process are counted towa | ecessarily enroll) to get the data and the total number of subjects Drop out, are screened out, etc.) |
| Total: | 80 | Of the total reques | ted indicate | Percent Male 0% | Percent Female 100% |
| | <b>4.1.1 Prov</b> i | de justification if a | l or more of one g | ender is targeted for par | ticipation |
| | Hysterecto | my | | | |
| <b>4.2.</b> How many subjects are needed to enroll to get the data sets required to answer the research question? For multi-center trials provide the number enrolled locally. | | | | | |
| Total: | 60 | | | | |
| 4.3 if | this is a m | ulti-center study, p | rovide the total nu | ımber of subjects to be e | nrolled from all centers: |
| Total: | n/a | | | | |
| 4.4 W | hich of the | following describe | the subjects (che | ck all that apply) | |
| ⊠ In <sub>l</sub> | patients | Outpatie | nts | Healthy volunteers | Condition-matched controls |
| 4.5 W | hat is the a | ge range of the sul | ojects? | | |
| Exact | Age Range | : 18 to 99 | See info | rmation below for requir | ed supplemental materials. |
| If age<br>includ | range<br>les | Required Supp | Required Supplemental Materials | | |
| 0-7 ye | ears | Parental conse | Parental consent form and Appendix Y required | | |
| 8-17 y | 8-17 years Child's assent, parental consent form and Appendix Y required | | | | |
| 4.6 List the criteria for subject INCLUSION in this study: | | | | | |
| ASA physical status I-III | | | | | |
| • Females >/=18-years of age | | | | | |
| <ul> <li>Scheduled for laparoscopic/robot-assisted hysterectomy.</li> </ul> | | | | | |

| 4.7 List the criteria for subject EXCLUSION from this study: | |
|---|---|
| Contraindication to surgical infiltra | tion or regional blockade |
| History of long term opioid intake | History of long term opioid intake (greater than 3 weeks prior to surgery) or chronic pain disorder |
| Inability to understand the informer | Inability to understand the informed consent and demands of the study |
| Surgery scheduled to start after 17 | 00 |
| 4.8 Are children included or excluded from | n this study? |
| Included – Appendix Y required – go | to question 4.8 |
| Excluded. Provide Justification below | v |
| No direct benefit to participation | (exclusion of children permissible) |
| Potential for direct benefit exists | for adults only (i.e. disease/condition does not occur in children) |
| Potential for direct benefit exists for children. Provide justification for exclusion of children: | |
| Note Regarding Exclusion of Children | |
| Note Regarding Exclusion of Children NIH guidelines advise that the exclusion be justified, so that potential for benefit is not unduly denied. Indicate whether there | |
| is potential for direct benefit to subjects in this study and if so, provide justification for excluding children. | |
| Note: If inclusion of children is justified, but children are not seen in the PI's practice, the sponsor must address plans to include children in the future or at other institutions. | |
| 4.9 Indicate if the research includes or specifically targets the populations listed below for participation. | |
| Inclusion of the populations below, either incidentally or by design, requires the investigator to provide additional information to the IRB. In some cases, such as the inclusion of prisoners, certification by the Office of Human Research Protection is required by federal regulations. If, after final approval, the subject population pool changes to include any listed below, complete a Change in Protocol Form and complete any relevant appendices. | |
| Population group/description | Resources and Required supplemental materials |
| Children | Appendix Y required. Review the University of Minnesota policy regarding Safety of Minors |
| Pregnant women/fetuses/neonates | Appendix B required. |
| | See guidance at <u>45CFR46 subpart B</u> and <u>http://www.research.umn.edu/irb/guidance/women.html.</u> |
| Prisoners | Appendix C required See guidance at 45 CFR 46 subpart C |

| Minority groups | Appendix I "Populations with Special Considerations" required. |
|---|---|
| Groups with socioeconomic or educational disadvantage | Appendix I "Populations with Special Considerations" required. |
| Non-English speakers targeted | Appendix I "Populations with Special Considerations" and consent forms in the language spoken by participants and an English translation. |
| Non-English speakers included (i.e., non-English speakers will not be turned away) | See guidance regarding the <u>short form consent process</u> . Consent short forms in Arabic, Croatian, French, Hmong, Khmer, Lao, Oromo, Russian, Somali, Spanish and Vietnamese are available for download. |
| Adults lacking capacity to consent and/or adults with diminished capacity to consent including, but not limited to, those with acute medical conditions, psychiatric disorders, neurologic disorders, developmental disorders and behavioral disorders. | Appendix I "Populations with Special Considerations" required. |

| Section 5 Study Location(s) | | |
|---|---|---|
| | Indicate in the table below all of the locations where the research will take place. | |
| | LOCATION | Required Supplemental Materials |
| $\boxtimes$ | Hospital/Clinic (specify below) | |
| | University of Minnesota Medical Center (UMMC) – | |
| | Fairview, Amplatz | |
| | Fairview Health Services (Southdale, Ridges, Lakes, | |
| | Northland | |
| | Gillette Children's Specialty Healthcare | |
| | Clinical and Translational Science Institute (CTSI) | |
| | University of Minnesota Physicians (UMP) Clinics | |
| | (Oncology Clinic, Phalen, Family Medicine, etc.) | |
| | Fairview Clinics (Maple Grove, Oxboro, Eden Center, | |
| | etc.) | |
| | TRIA Orthopedic Center | |
| | Other, Specify: | |
| | University Campus (Non-clinical location) | |
| | Minneapolis/St Paul Rochester | |
| | Duluth Crookston | |
| | Morris | |
| | Other, specify: | |
| | Veteran's Administration Medical Center | Veteran Administration IRB approval |

| | Center for Magnetic Resonance Research (CMRR) | Submit Documentation of CMRR Safety Committee approval. |
|---|---|---|
| | | CMRR users must submit the completed CMRR Device and Safety Review form to the CMRR prior to submission of their IRB application. A draft copy of the IRB application must be included for CMRR Safety Committee review. Documentation of approval by the CMRR Safety Committee will be provided to the researcher to include with the IRB application. |
| | Elementary school/secondary school | Submit Appendix M "Research in Schools" and appropriate documentation of approval from school district |
| | University of Minnesota Child Care Center | |
| | Prison/Halfway House | Submit Appendix C "Prisoners as Subjects" |
| | Federal Prison State Prison Halfway house, specify: | |
| П | International Location | Submit Appendix K "International Research" |
| | Sovereign Nation within United States borders | Submit documentation of approval from sovereign nation |
| | Military base or facility owned by any component of the<br>Department of Defense | Submit Appendix D "Department of Defense" |
| | Nursing home, specify: | Documentation of approval from site administrators |
| | Community center, specify: | Documentation of approval from site administrators |
| | Research will be conducted online | |
| | Other, specify: | |
| Sect | ion 6 Recruitment & Compensation | |
| University of Minnesota policy prohibits researchers from accepting gifts for research activities. Research staff must decline any incentive (i.e. finders fees, recruitment bonus, etc.) offered by the study sponsor connected with subject enrollment or completion of the research study. For more information, please see Code of Conduct | | |
| | //www1.umn.edu/regents/policies/academic/Code of Condu<br>Which of the statements below describes the recruitment stra | |
| 6.1 V | vnich of the statements below describes the recruitment stra | ategy? If both apply, select both. |
| | Statement A. Potential subjects will self-identify based on re respondent driven sampling. <b>If ONLY statement A selected,</b> | |
| | Statement B. Potential subjects will be recruited based on in (medical records, student records). This also includes subject | |

| patient population. If statement B is selected, answer the question | ns 6.1.1. – 6.1.3 below |
|---|---|
| 6.1.1 Explain how the researcher has legitima | |
| The PI is a surgeon at the University of Minnesota | |
| 6.1.2 Identify who will make initial contact wi | th potential subjects. |
| THe PI or Co-Investigators | |
| 6.1.3 Will the records include MEDICAL record | ds? |
| No, go to question 6.2 | |
| Yes. Indicate the mechanism the PI will use to confirm that the patient has agreed to release their PHI contained in their medical record for research purposes; for example, the patient has documented consent to research on their treatment, intake or hospital admitting form. (MN Statue 144.334 Subd. 3; Access to Medical Records for Research) | |
| Academic Health Center Information | Exchange (AHC-IE) |
| Other. Describe: EPIC | |
| Check the box(es) that describe the recruitment nitted with this application. | t strategy. Any required documents as detailed below should be |
| Method | Required Supplemental Materials |
| Flyers | Submit Flyer with application |
| Newspaper ads | Submit draft of ad with application |
| Radio or television ads | Submit script with application |
| Social networking sites | Text, page mock up or description of posting including any images or videos |
| | Indicate site(s): |
| Letters or emails | Submit letter or email with application |
| Phone call | Submit phone script with application |
| Group presentations | Submit outline of presentation and any materials provided to participants with application |
| University of Minnesota research recruitment tool (e.g. REP, SONA or Carlson School Recruitment) | |

| | Non-University of Minnesota research recruitment tool (e.g. MTURK, Research Match) | |
|---|---|---|
| | Other method not described above | Specify: Patients will be identified in clinic. There they will be presented with the consent form and then on day of surgery they will sign final consent after speaking with the anesthesiologist. |
| | rovide a brief narrative to describe the recruitn<br>be informed of the research. | nent process. Include in the description how potential subjects |
| they<br>as w | will sign final consent after speaking with the an | e presented with the consent form and then on day of surgery lesthesiologist. They will be able to ask quesitons in surgery clinic II be made available so they can ask questions regarding the |
| | | nent, services without charge or extra credit be provided to the |
| subje | ect for participation in research? | d Daire as |
| | No If no, go to Section 7 Confidentiality and | d Privacy |
| | Yes Complete 6.4.1 – 6.4.4 | |
| | 6.4.1 Indicate the type of compensation and this/her participation. | he maximum value a subject may receive during the course of |
| | 6.4.2 When will compensation be provided? I prorated and the compensation schedule | Include in the response if payment for multiple visits is |
| | 6.4.3 Who will receive the compensation? | |
| | Subject | |
| | Other, specify: | |
| | 6.4.4 Will Research Experience Points (REP) b | e awarded? |
| | Yes | |
| | □ No | |

# Section 7 Confidentiality and Privacy

| <b>Confidentiality</b> refers to how the subject's identifiable data will be handled, managed, stored, and, if applicable, disseminated. | | | | | | |
|---|---|---|---|---|---|---|
| | - | rs to having con<br>ally) with others | | er the extent, timi | ing, and | circumstances of sharing oneself (physically, behaviorally |
| 7.1. | Will res | earchers mainta | ain any | / identifiers (e.g. n | names, | addresses, telephone numbers, etc.)? |
| | No. G | o to question 7. | 13 | | | |
| | Yes. | | | | | |
| 7.2 l | ndicate | which of the di | rect id | entifiers below wi | ill be m | aintained? |
| | ☐ Fu | ull names | | Initials | | Photographs of participant |
| | | elephone<br>umbers | | Email address | | Videos of participant |
| | Ві | irth date | | Postal Address | | Other: |
| 7.3 Why it is necessary to maintain direct identifiers? | | | | | | |
| 7.4 Describe the coding system that will be used to protect against disclosure of these identifiers. | | | | | | |
| 7.5 How long will the link between identifiers and code be maintained? | | | | | | |
| 7.6 Could any disclosure of the participant's responses place the participant at risk of criminal or civil liability or could the disclosure be damaging to the participant's financial standing, employability, or reputation? | | | | | | |
| | No | | | | | |
| | Yes Explain how the researcher will mitigate these risks (e.g. limiting access to identifiers, obtaining a Certificate of Confidentiality, etc.)? | | | | | |
| 7.7 V | Vill the | researcher obta | nin a <u>C</u> | ertificate of Confi | dentiali | ty for this project? |
| No | | | | | | |
| | Yes | Documentation | n of Ce | ertificate of Confid | entialit | y must be provided to the IRB when obtained. |

| 7.8 How long will the identifiable data be maintained? |
|---|
| n/a |
| 7.9 What format will be used to maintain the data (paper, digital, electronic media, video, audio or photographic)? |
| n/a |
| 7.10 Where will data be stored? |
| All data will be stored on a password protected encrypted jump drive in a locked drawer in locked office. |
| 7.11 What security provisions will be taken to protect the data (password protection, encryption, etc.)? See the University of Minnesota's <a href="Safe Computing recommendations">Safe Computing recommendations</a> |
| password protection and encryption |
| 7.12 Will a copy of the consent form or other research study information be placed in the subjects' non-research records such as medical, employment or educational records? |
| No |
| Yes This information must be included the confidentiality section of the consent form. |
| 7.13 Even if direct identifiers are not recorded or maintained, are there potential ethical or legal circumstances when it would be necessary to break confidentiality (e.g. requirements for mandated reporting)? |
| No |
| Yes This information must be included in the consent form. <b>Explain below the circumstances when breaking confidentiality is required.</b> |
| 7.14 Describe the conditions under which interaction with subjects will occur (e.g., consent discussion occurs in a private room). Explain how these conditions adequately protect the PRIVACY interests of subjects. |
| consent discussion will occur in a private room as well as signing of the consent. All staff will undergo research training to ensure they protect privacy of the patients. |

#### 

Federal criteria for risk assessment make some studies eligible for Expedited Review (see 45 CFR46.110 and 21 CFR 56.110). Expedited review categories are below and may also be found at <a href="http://www.irb.umn.edu/expedited.html">http://www.irb.umn.edu/expedited.html</a>

Studies eligible for Expedited Review must meet the federal definition of minimal risk which is:

The probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological

| examinations or tests. | | |
|---|---|---|
| 8.1 W | hat is | the level of risk to subjects in this research study? |
| | Great | er than minimal risk (full committee review required) – go to Section 9 Informed Consent Process |
| | Not g | reater than minimal risk. |
| | | w the table in question 8.2 below and check the box next to the expedited review category the igator asserts applies to this research. |
| | | Final expedited review eligibility decisions are made by the IRB after initial review of the application. is involving drugs/biologics or devices are rarely eligible for expedited review. |
| | | e box next to the Expedited Review Categories (2-7) that apply to the proposed project. Per UMN IRB cal studies involving drugs or devices are not eligible for expedited review category 1. |
| Not | | 1. Clinical studies of drugs and medical devices only when condition (1) or (2) is met. |
| availab<br>per UN<br>IRB pol | ΛN | <ol> <li>Research on drugs for which an investigational new drug application (21 CFR Part 312) is not required.</li> <li>(Note: Research on marketed drugs that significantly increases the risks or decreases the acceptability of the risks associated with the use of the product is not eligible for expedited review.)</li> </ol> |
| | | <ol> <li>Research on medical devices for which (i) an investigational device exemption application (21 CFR Part<br/>812) is not required; or (ii) the medical device is cleared/approved for marketing and the medical device<br/>is being used in accordance with its cleared/approved labeling.</li> </ol> |
| | Cat. 2 | Collection of blood samples by finger stick, heel stick, ear stick, or venipuncture as follows: |
| | | 1. from healthy, nonpregnant adults who weigh at least 110 pounds. For these subjects, the amounts drawn may not exceed 550 ml in an 8 week period and collection may not occur more frequently than 2 times |
| | | per week; or |
| | | 2. from other adults and children, considering the age, weight, and health of the subjects, the collection procedure, the amount of blood to be collected, and the frequency with which it will be collected. For |
| | | these subjects, the amount drawn may not exceed the lesser of 50 ml or 3 ml per kg in an 8 week period and collection may not occur more frequently than 2 times per week. |
| | Ca+ 2 | Prospective collection of biological specimens for research purposes by noninvasive means. |
| | Cat. 3 | Examples: |
| | | 1. hair and nail clippings in a nondisfiguring manner; |
| | | <ol> <li>deciduous teeth at time of exfoliation or if routine patient care indicates a need for extraction;</li> <li>permanent teeth if routine patient care indicates a need for extraction;</li> </ol> |
| | | 4. excreta and external secretions (including sweat); |
| | | 5. uncannulated saliva collected either in an unstimulated fashion or stimulated by chewing gumbase or |
| | | wax or by applying a dilute citric solution to the tongue; |
| | | 6. placenta removed at delivery; |
| | | 7. amniotic fluid obtained at the time of rupture of the membrane prior to or during labor; |
| | | 8. supra- and subgingival dental plaque and calculus, provided the collection procedure is not more invasive than routine prophylactic scaling of the teeth and the process is accomplished in accordance with |
| | | accepted prophylactic techniques; |
| | | <ol> <li>mucosal and skin cells collected by buccal scraping or swab, skin swab, or mouth washings;</li> <li>sputum collected after saline mist nebulization.</li> </ol> |
| | _ | Collection of data through noninvasive procedures (not involving general anesthesia or sedation) routinely |
| | Cat. 4 | employed in clinical practice, excluding procedures involving x-rays or microwaves. |
| | | Where medical devices are employed, they must be cleared/approved for marketing. (Studies intended to |
| | | evaluate the safety and effectiveness of the medical device are not generally eligible for expedited review, |

including studies of cleared medical devices for new indications.) Examples: 1. physical sensors that are applied either to the surface of the body or at a distance and do not involve input of significant amounts of energy into the subject or an invasion of the subject's privacy; 2. weighing or testing sensory acuity; 3. magnetic resonance imaging; 4. electrocardiography, electroencephalography, thermography, detection of naturally occurring radioactivity, electroretinography, ultrasound, diagnostic infrared imaging, doppler blood flow, and echocardiography; 5. moderate exercise, muscular strength testing, body composition assessment, and flexibility testing where appropriate given the age, weight, and health of the individual. Research involving materials (data, documents, records, or specimens) that have been collected, or will be Cat. 5 collected solely for nonresearch purposes (such as medical treatment or diagnosis). (NOTE: Some research in this category may be exempt from the HHS regulations for the protection of human subjects. 45 CFR 46.101(b)(4). This listing refers only to research that is not exempt.) Cat. 6 Collection of data from voice, video, digital, or image recordings made for research purposes. Cat. 7 Research on individual or group characteristics or behavior (including, but not limited to, research on perception, cognition, motivation, identity, language, communication, cultural beliefs or practices, and social behavior) or research employing survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies. (NOTE: Some research in this category may be exempt from the HHS regulations for the protection of human subjects. 45 CFR 46.101(b)(2) and (b)(3). This listing refers only to research that is not exempt.)

### **Section 9 Informed Consent Process**

### **Document the Elements of the Informed Consent Process**

It is the responsibility of the investigator to assess comprehension of the risks and benefits of participation in the research and only enroll subjects who can demonstrate understanding of the research study (45 CFR 46.116). The federal regulations require that consent be in language understandable to the subject. If subjects do not comprehend English, translated consent forms are required, or the use of short forms with an oral explanation can be accepted.

Consent forms must be submitted for IRB review. It is highly recommended that researchers use the sample consent for template available on the <u>IRB Forms page</u>. Do not submit sponsor prepared forms without editing the form to include University of Minnesota IRB standard language and all essential elements of informed consent.

Resources for preparing consent forms are available at:

<u>Informed Consent Online Tutorial</u> – <a href="http://www.research.umn.edu/consent/">http://www.research.umn.edu/consent/</a>

If the researcher is requesting a waiver of consent, complete questions 9.9 and 9.10 only. Be advised that waiver of consent is rarely granted.

**9.1 Document the informed consent process timeline.** Detail when consent will be discussed and documented in relation to research data collection, if there will be any waiting period or if process will occur over multiple contacts or clinical visits.

The consent will be discussed in the ciinic visit with the surgeon. They will be given a copy of the consent and a phone number to call if they have questions. Then on the day of surgery after they have had adequate time to

| revie | review the consent they will sign consent after discussion with the anesthesiologist (co-PI). | |
|---|---|---|
| <b>9.2 Will anyone not listed on this application obtain consent?</b> Except in rare circumstances, all individuals who will obtain consent must be listed as research personnel on the IRB application so that basic human subjects' research training is documented. If in-person consent will not be obtained, select the option below and provide rationale. | | |
| $\boxtimes$ | No | If no, go to question 9.3 |
| | Yes | Explain who, other than those listed as personnel on this application, will obtain consent |
| | N/A | In-person consent will not be obtained. Explain below: |
| | | a brief description of the plan to train those individuals who will be obtaining consent from subjects to n this project. |
| | | complete CITI training. |
| | - | one obtaining consent must complete <u>CITI training</u> . |
| 9.4 V | Vill all | subjects consent for themselves? |
| | Yes | If yes, adults lacking capacity to consent must be listed in the exclusion criteria (question 4.7). |
| | No | If no, indicate below who, when appropriate, will provide consent |
| | | Parent/guardian |
| | | Legally authorized representative – Appendix I required |
| | - | uestions will be asked to assess the subjects' understanding? Questions should be open-ended and go uiring a yes/no response. |
| What | are th | e benefits and risks of the tap or infiltration? |
| What | What are the benefits and risks of either local anesthetic medication? | |
| How will your pain be managed post-operatively in both options of the study? | | |
| What are the alternative treatment options to control your pain post-operatively? | | |
| What | will be | done if you have an allergic reaction or reaction to the pain medication in this study? |
| 9.6 Participation in research must be voluntary. Describe the steps taken to minimize the possibility of undue influence on potential subjects. | | |
| As the intervention we are providing two options which is the current standard of care, it is considered safe and efficacious. We will discuss the options, as well as the risks and benefits with the patient. No additional benefit is gained by the anesthesiologist if this technique is used and this will be discussed with the patient. | | |
| | | ects in Case of Accident |
| If this research involves a potential for injury, injury compensation language must be included in the consent form (see | | |
| 21 CFR 50.25). If a contract to pay for research-related injuries exists, the language in the consent form should not contradict the language in the contract. | | |
| 9.7 | s there | a potential for research related injury? |

| ☐ No | If no, go to question 9.8 |
|---|---|
| Yes | If yes, indicate which of the following statements is included in the consent form |
| | Non-Sponsor Funded Compensation |
| | Then spensor runded compensation |
| | In the event that this research activity results in an injury, treatment will be available, including |
| | first aid, emergency treatment and follow-up care as needed. Care for such injuries will be billed |
| | in the ordinary manner, to you or your insurance company. If you think that you have suffered a |
| | research related injury let the study physicians know right away. |
| | research related injury let the study physicians know right away. |
| | Sponsor Funded Compensation |
| | In the event that this research activity results in an injury, treatment will be available, including |
| | In the event that this research activity results in an injury, treatment will be available, including |
| | first aid, emergency treatment and follow-up care as needed. Care for such injuries will be billed in the ordinary manner, to you or your insurance company. The sponsor of the study has some |
| | funds available to pay for care for injuries resulting directly from being in this study. If you think |
| | that you have suffered a research related injury and that you may be eligible for reimbursement |
| | of some medical care costs, let the study physicians know right away. |
| | of some medical care costs, let the study physicians know right away. |
| | If the preferred injury compensation language is unacceptable to the study sponsor, the |
| | following alternative language may be used: |
| | Under some circumstances the sponsor of the study will pay for care for injuries resulting directly |
| | from being in the study. If you want information about those circumstances or if you think you |
| | have suffered a research related injury let the study physicians know right away. |
| Waiving Do | cumentation of Consent |
| Waiving wr | itten documentation assumes that there will be an informed consent process but signatures will not be |
| collected or | the consent form. The IRB may waive the requirement for written documentation under specific |
| conditions. | |
| 9.8 Does th | e researcher wish to waive documentation of consent? |
| No No | If no, go to question 9.9 |
| Yes | If yes, check the statement below that applies to justify waiving documentation of consent. If neither |
| | statement applies, researcher may not request waiver of documentation |
| | The only record linking the subject and the research would be the consent form and the principal |
| | risk of the research would be the potential harm from a breach of confidentiality (the IRB may |
| | allow an option to sign or decline) |
| | The research presents no more than minimal risk and includes no procedures for which written |
| | consent is normally required outside the research context. |
| NOTE: Rese | archers requesting a waiver of documentation must submit a consent form without signature lines with |
| the IRB app | · |
| PP | |
| Waiving Co | nsent |
| _ | y, in some rare and specific circumstances, waive the requirement for consent in accordance with 45 CFR |
| | Answer the guestions below to determine if waiver of consent may be considered. |

| 9.9 Does th | e researcher wish to waive consent? | |
|---|---|---|
| No Yes | | |
| Section 1 | 0 Funding | |
| 10.1 Has funding for this project been applied for, requested or received or do you intend to request/apply for funding? | | |
| □ No | Explain how the research will be conducted w | ithout funding: |
| | Indicate in the table below who will provide/ma | anage funds. |
| Funds pro- | ided/managed by | Poguired Supplemental Materials |
| Funds provided/managed by Internal University of Minnesota (departmental | | Required Supplemental Materials none |
| | , internal grant program, etc.) | Tione |
| | Describe: Anesthesiology funds | |
| | rsity of Minnesota Sponsored Project Funding | Appendix A required |
| | Jniversity of Minnesota source or management | Appendix A required |

## **Section 11 Conflict of Interest**

Federal Guidelines emphasize the importance of assuring there are no conflicts of interest in research projects that could affect the welfare of human subjects. Reporting of financial interests is required from all individuals responsible for the design, conduct or reporting of the research. If this study involves or presents a potential conflict of interest, additional information will need to be provided to the IRB.

Examples of conflicts of interest may include, but are not limited to:

• A researcher participating in research on a technology, process or product owned by a business in which the researcher or family member holds a significant financial interest or a business interest.

- A researcher participating in research on a technology, process or product developed by that researcher or family member.
- A researcher or family member assuming an executive position in a business engaged in commercial or research activities related to the researcher's University responsibilities.
- A researcher or family member serving on the Board of Directors of a business from which that member receives University supervised Sponsored Research Support.
- A researcher receiving consulting income from a business that funds his or her research.
- A researcher receiving consulting income from a business that could benefit from the results of research sponsored by a federal agency (i.e. NIH).

| | federal agency (i.e. NIH). |
|---|---|
| intere<br>resea | Do any of the Investigators or personnel listed on this research project have a business interest or a financial est of \$10,000 or more (\$5,000 or more if research is funded by a Public Health Service (PHS) agency or rcher is involved in clinical health care) associated with this study when aggregated for themselves and their y members? |
| | No |
| $\boxtimes$ | Yes List the investigator(s) with conflicts: |
| | Jacob Hutchins is on speakers bureau, consultant and has received research funds |
| | Do any of the investigators or personnel (when aggregated for themselves and their family members) listed is research have: |
| | 11.2.1 Ownership interests more than \$10,000 (\$5,000 if research is funded by PHS or researcher is involved in clinical health care) when the value of interest could be affected by the outcome of the research? |
| | No |
| | Yes List the investigator(s) with conflicts: |
| | 1.2.2 Ownership interests exceeding 5% interest in any one single entity (or any equity interest in a non-publicly traded entity if research is funded by PHS or researcher is involved in clinical health care)? |
| | No No |
| | Yes List the investigator(s) with conflicts: |
| | 11.2.3 Compensation greater than \$10,000 (\$5,000 if research is funded by PHS or researcher is involved in clinical health care) when the value of the compensation could be affected by the outcome of the research? |
| | ⊠ No |
| | Yes List the investigator(s) with conflicts: |

| 11.3 Have all business or financial interests indicated above been reported? |
|---|
| □ No |
| N/A There are no conflicts of interest on this study |
| <ul> <li>University of Minnesota researchers need to report business or financial interest online via the <u>Report of External Professional Activities (REPA)</u></li> </ul> |
| <ul> <li>Fairview Health System researchers need to complete the <u>Fairview Health Services Conflict of Interest Disclosure</u> <u>forms</u> and submit the completed forms to the Fairview Office of Research.</li> </ul> |
| <ul> <li>Gillette Children's Specialty Healthcare researchers must contact the Director of Research Administration, at<br/>651-229-1745.</li> </ul> |
| The IRB will verify that a management plan is in place with the Conflict of Interest (COI) Program. If the COI Program does not have an approved management plan in place for this research, they will contact the individual(s) for additional information. |
| Final IRB approval cannot be granted until the IRB has reviewed the management plan and all potential conflict matters are settled. The IRB receives a recommendation from the Conflict of Interest Review Committee regarding disclosure to subjects and management of any identified conflict. The convened IRB determines what disclosure language should be in the consent form. |
| Section 12 Research Services, Assessment and Oversight |
| Section 12.1 RESEARCH COLLABORATIONS |
| 12. 1 Does this research project involve collaborations with any sites or personnel outside of the University of Minnesota, its coordinate campuses, the Fairview Health Systems or Gillette Children's Specialty Healthcare? |
| No Go to question section 12.2 |
| Yes Briefly describe the collaboration (with whom and for what purpose): |
| Additional requirements for ensuring appropriate IRB oversight may apply. These requirements are often dependent on whether or not the site/personnel is considered "engaged" in human subjects research according to federal definitions. Contact the UMN IRB office ( <a href="mailto:irb@umn.edu">irb@umn.edu</a> ) to determine how IRB oversight of the research activity with the external site/personnel should be address. |
| Section 12.2 AFFILIATED ENTITIES WITH OVERSIGHT RESPONSIBILITIES |
| 12.2.1 Will this research use services, resources, or funding from the Clinical and Translational Science Institute? Examples include pilot funding, career development awards, biostatistics support, facilities, staffing, project management, regulatory assistance, or informatics consultation and support |
| No Go to question 12.2.2 |

| Yes | Provide CTR Portal ID#: |
|---|---|
| 12.2.2 Doe | es this research require Masonic Cancer Center Protocol Review Committee (CPRC) review? |
| | required to evaluate, approve or reject, monitor, and re-review on an annual basis all University of Minnesota<br>cer research protocols including those with non-therapeutic intent. |
| ⊠ No | Go to question 12.2.3 |
| Yes | Documentation of approval must be provided to receive final IRB approval. |
| 12.2.3 Wi | Il this research utilize Gillette Children's Specialty Healthcare resources or medical records? |
| ⊠ No | Go to section 12.3 |
| Yes | If using Gillette resources, please contact: |
| | Joyce Trost, PT<br>Research Administration Manager |
| | Gillette Children's Specialty Healthcare 651-325-2339/651-312-3182/jtrost@gillettechildrens.com |
| | Il this research use Magnetic Resonance (MR) Devices housed at the Center for Magnetic Resonance CMRR) facilities? |
| ⊠ No | Go to section 12.3 |
| Yes | Review and approval by the CMRR Safety Committee is required prior to IRB submission. |
| | CMRR users must submit the completed CMRR Device and Safety Review form to the CMRR prior to submission of their IRB application. A draft copy of the IRB application must be included along with the CMRR Device and Safety Review form for CMRR Safety Committee review. Documentation of approval by the CMRR Safety Committee will be provided to the researcher to include with the IRB application submission. |
| Section | 12.3 PAYMENT FOR RESEARCH RELATED SERVICES |
| | es the protocol require the use of tests, procedures, clinic space, clinic visits, professional fees, lab harmacy services, or hospital services in order to answer the research question? |
| ☐ No | Go to section 12.4 |
| Yes | |
| 12.3.2 Wil | I subjects or a third party be charged for research related procedures? |
| No | |
| ⊠ Yes | <b>Explain:</b> These are standard of care and as such are charged to the patient as per routine |
| | Provide written documentation from the FDA to charge for investigational products. |

| 12.3.3 Will Services be provided by Fairview Health Service or U of M Physicians? |
|---|
| □ No |
| Yes Provide TASCS Number: |
| Provide a copy of the TASCS billing grid noting whether the study does or does not meet Medicare criteria for a Qualifying Clinical Trial. |
| Applications will not be assigned for review until the TASCS information is submitted. |
| CLINICALTRIALS.GOV REGISTRATION |
| Important Information about clinicaltrials.gov registration |
| Resources available, penalties for failure to register and publication requirements |
| Potential risks associated with failure to register with clinicaltrials.gov: |
| Loss of funding (National Institute of Health) |
| Financial penalty levied against the PI |
| Denial of publication (ICMJE) |
| Denial of payment to healthcare providers. |
| Section 801 of the Food and Drug Administration Amendments Act (FDAAA 801) establishes penalties for Responsible Parties who fail to comply with registration or results submission requirements. Penalties include civil monetary penalties and, for federally funded studies, the withholding of grant funds. |
| The International Committee of Medical Journal Editors (ICMJE) defines a clinical trial as any research project that prospectively assigns human subjects to intervention or concurrent comparison or control groups to study the cause-and-effect relationship between a medical intervention and a health outcome. Medical interventions include drugs, surgical procedures, devices, behavioral treatments, process-of-care changes, and the like. |
| Research projects that meet the ICMJE definition may not be accepted for publication if they are not registered in a registry that is electronically searchable and accessible to the public at no charge. For more information on this requirement see <a href="http://www.icmje.org">http://www.icmje.org</a> Note that retrospective registration of projects is not allowed. |
| Additionally, healthcare providers are required to include the clinicaltrials.gov number on all claims during the time period the patient participates in the study. |
| The Clinical and Translational Science Institute (CTSI) will assist University of Minnesota investigators to comply with the registration requirement. Complete the section below to document status or determine if registration is required. Applications submitted without a Clinicaltrials.gov registration number (either received or pending) will be forwarded to the CTSI for review. |
| Section 12.4 CLINICALTRIALS.GOV REGISTRATION DETERMINATION |
| 12.4.1 Is this project registered with clinicaltrials.gov? |

Go to 12.4.2

☐ No

| Xes | Clinicaltrials.gov registration number:pending | |
|---|---|---|
| | If registration is pending enter "pending" in the space provided. | |
| Doos this pro | Section complete. Go to Section 12.5 rject meet the Food and Drug Administration Amendments Act ( | EDAAA) definition of "applicable |
| • | ? Applicable clinical trials generally include controlled, clinical ir | • • |
| | ed trials of devices that include health outcomes, including pedia | |
| and controlle | that that of devices that melade health outcomes, melading peak | active postition received and vehicles. |
| 12.4.2 Is regi | stration with clinicaltrials.gov required? | |
| No | The PI understands the registration requirements and the co | nsequences, as described above, of |
| | failure to register if applicable. CTSI will review this application | - |
| | decision. CTSI will contact the PI and the IRB to confirm regist | ration requirement. If registration is |
| | required, the PI may request assistance with this process from | |
| Unsure | CTSI will contact the PI and the IRB with a determination reg | |
| | registration is required, the PI may request assistance with the 12.5 | nis process from CTSI. Go to Section |
| Yes | Answer the questions below to determine who (either the PI | or other entity) is responsible for |
| | registration with clinicaltrials.gov | |
| | Is this study initiated by a University of Minnesota | No |
| | investigator? | Yes – registration by PI required. |
| | Is this study federally sponsored and the University of | No |
| | Minnesota is the only study site OR the study's coordinating | Vos registration by DI required |
| | center? | Yes – registration by PI required. |
| | Is a University of Minnesota investigator the holder of an | ⊠ No |
| | Investigational New Drug (IND) application for the test | _ |
| | article OR it has been determined the proposed use of the Yes – registration by PI required. | |
| | test article is IND exempt? | 5-7 |
| | Is a University of Minnesota investigator the holder of an | ⊠No |
| | Investigational Device Exemption (IDE) for the device being | |
| | studied OR a non-significant risk (NSR) determination has been made for the device being studied? | Yes – registration by PI required. |
| | | royidad hafara final IPR approval is |
| | If registration is required, the registration number must be p | |
| | granted. Email <a href="mailto:ctsi@umn.edu">ctsi@umn.edu</a> for additional information and registration assistance. CTSI will evaluate all applications not registered with clinicaltrials.gov. | |
| | evaluate an approacions not registered with chimeantialsigor | • |
| Section 12 | 2.5 SCIENTIFIC ASSESSMENT | |
| Research inv | olving human subjects must be reviewed for sound scientific de | sign prior to review by the IRB |
| committee. | Documentation of scientific assessment including the content o | f the review must be provided before the |
| project will be reviewed by the IRB. Scientific assessment is not required for new studies that meet the federal | | |
| criteria for ex | spedited review. If a study is submitted for expedited review bu | t is determined by the IRB to NOT meet |

the criteria for expedited review, then scientific peer review will be required before IRB review.

review eligible. GO TO Section 13 Additional Staff.

Project qualifies for expedited review. Sections 12.5, 12.6 and 12.7 are not required if expedited

N/A

12.5.1 Has the IRB scientific assessment requirement been met?

| ⊠ Yes | Indicate below<br>met | how the requirement has been | Required supplemental materials |
|---|---|---|---|
| | Option1 | Reviewed by a <b>federal funding</b> | |
| | | agency (National Institutes of | |
| | | Health, National Science | |
| | | Foundation, etc.) employing peer | |
| | | review mechanisms for awarding | |
| | | of funding. | |
| | Option 2 | Reviewed by a nationally based | |
| | | non-federal funding agency | |
| | | (March of Dimes, American | Note: industry-sponsored clinical trials designed |
| | | Academy of Pediatrics, etc.) | by the sponsor with or without external |
| | | employing peer review | consultants do not satisfy this criterion for |
| | | mechanisms for awarding of | independent peer-review. |
| | Option 3 | funding Reviewed by <b>locally constituted</b> | Attach the review and the signed form |
| | | mechanisms using peer review | Attach the review and the signed form documenting that departmental or collegiate |
| | | for awarding of funding, or for | peer review of the research protocol has been |
| | | permission to use resources: | performed. |
| | | Cancer Protocol Review | periori in car |
| | | Committee (CPRC); CTSI funded | |
| | | pilot awards; Vikings; | |
| | | departmental peer review etc. | |
| | Option 4 | Reviewed by HRPP facilitated | Submit approval notification with application. |
| | | Scientific Assessment committee | |
| Section 12. | 6 DATA AND | SAFETY MONITORING PLA | N |
| A data and saf | ety monitoring p | olan (DSMP) is meant to assure that | each clinical investigation has a system for |
| oversight and | monitoring of th | ne conduct of the clinical investigatio | n. This oversight is intended to ensure the safety |
| of the particip | ants and the val | idity and integrity of the data. A DSN | MP should be commensurate with the risks. |
| A DSMP can b | e as simple as th | e investigator reporting adverse eve | nt information to the IRB. A DSMP can be as |
| | | Safety Monitoring Board. | |
| · | J | , | |
| A DSMP can in | iclude clinical tri | al monitoring. Clinical trial monitori | ng refers to the methods used to oversee the |
| conduct of, an | d reporting of d | ata from, clinical investigations inclu | ding appropriate clinical investigator supervision of |
| study site staf | f. Monitoring act | tivities include communication with | the investigator and the study site staff; review of |
| the study site' | s processes, pro | cedures, and records; and verificatio | n of the accuracy of the data. |
| 12.6.1 In addi | tion to the Princ | cipal Investigator, are there other DA | ATA monitoring entities responsible for this |
| | ect all that apply | • | |
| = | | itity monitoring DATA. | |
| Yes | A review en | itity will provide ongoing DATA mor | nitoring |
| | | d T | CTCI) |
| Clinical and Translational Science Institute (CTSI) Data coordinating center or project principal investigator (multi-center studies) | | | |
| | Commercial sponsor, contract research organization (CRO) | | |

| Other: | | | | | |
|---|---|---|---|---|---|
| Other: 12.6.2 In addition to the Principal Investigator, are there other SAFETY monitoring entities responsible for this function? Select all that apply. No, the PI is the only entity monitoring SAFETY. Yes Select all below that apply A Data Safety Monitoring Board (DSMB) will be appointed. When established, the list of the DSMB members including their affiliation and credentials and the DSMB charter must be submitted to the IRB. A description of the DSMB must be provided with the | | | | | |
| | application. A Data and Safety Monitoring Board (DSMB) is an independent group of experts that advises the study investigators. Primary responsibilities of a DSMB are to 1) periodically review and evaluate the accumulated study data for participant safety, study conduct and progress, and, when appropriate, efficacy, and 2) make recommendations concerning the continuation, modification, or termination of the trial. The DSMB considers study-specific data as well as relevant background knowledge about the disease, test agent, or patient population under study. The DSMB reports should be provided to the IRB as they are received. Medical Monitor Cancer Center Data Safety Monitoring Council Other, describe: | | | | |
| Section 12. 7 DATA AND SAFETY MONITORING RESPONSIBILITIES | | | | | |
| Data to be m | onitored | PI | Review entity | DSMB/other | Unassigned |
| | (e.g., collection, reporting, and confidence of AEs, SAEs, and other study | | | | |
| Data Accuracy & Quality Assurance (e.g., data | | | | | |
| Trial Management (e.g., site coordination, enrollment and population distribution). | | | | | |
| Regulatory Issues (e.g., SAE reporting, IRB Actions, disclosures of conflict of interest). | | | | | |

## **Section 13 Additional Research Staff**

# **Co-Investigators**

Interim Analysis.

justification:

Co-Investigators, responsible for knowing and following the protocol, should be listed below. Include any individual who will have responsibility for the consent process, direct data collection from subjects, or follow-up.

It is the investigator's opinion that this protocol does not require a data safety monitoring plan. Provide

Note: If emailing this application to the IRB, all co-investigators must be cc'ed on the submission email.

| Co-Investigator Name (Last name, First name MI): | | | Highest Earned Degree: | |
|---|---|---|---|---|
| Argenta, Peter, | | | MD | |
| Affiliation and contact inform | nation | ' | | |
| ☐ University of Minnesota (complete contact info section 1 only) | | | ☐ Gillette (complete contact info section 2 only) | |
| ☐ Fairview (complete contact | info section 2 only) | Othe | er (complete c | ontact info section 2 only) |
| Required Contact information | U of M Internet ID (x.500): | argenta | | |
| Section 1 - U of M only | U of M Employee/student<br>ID Number: | | | |
| | University Department: | Department of Obstetrics, Gynecology and Women's Health, Division of Gynecologic Oncology | | |
| Required contact information | Address: | | Phone num | ıber: |
| Section 2 Non-U of M only | | | | |
| | | ☐Mobile ☐ Pager ☐Office Email address: | | |
| Occupational Position: | | | | |
| Faculty Physician Sta | ff Student Other: | | | |
| Project responsibilities: | | | | |
| Obtain consent from subjects | Provide access to patient pop | oulation 🔲 O | ther: | |
| Conflict of Interest: | | | | |
| Does this person have a reportabl | e conflict as defined in Section 13 | 1 of the applic | cation? | |
| ☐ Yes ⊠ No | | | | |
| Required CITI Human Subje | | | | HIPAA TRAINING |
| Date CITI completed (either in | itial or refresher course): | | | Check box below if HIPAA training is required. |
| Note: The IDD was in a second as | | MIPAA Required – Data contains R | | HIPAA Required – Data contains PHI |
| Note: The IRB requires researcher completion of initial course. For | | | | HIPAA Training completed through: |
| • | | • | | ☐ UMN |
| | | | | Other: |
| Signature/Digital signature/x.500 of Co-PI | | | Title of Co-PI | |
| Co-Investigator Name (Last name, First name MI): Highest Earned Degree: | | | | |
| Hutchins, Jacob | | | MD | |
| Affiliation and contact information | | | | |
| University of Minnesota (complete contact info section 1 Gillette (complete contact info section 2 only) | | | | |
| Fairview (complete contact | info section 2 only) | Othe | er (complete c | ontact info section 2 only) |

| Required Contact information | U of M Internet ID (x.500): | hutc0079 | | |
|---|---|---|---|---|
| Section 1 - U of M only | U of M Employee/student ID Number: | 2182198 | | |
| | TD Number. | | | |
| | University Department: | Anesthesiology | | |
| Required contact information | Address: | | Phone nu | mber: |
| Section 2 Non-U of M only | | | | Пр Пост |
| | | | ☐ Mobile ☐ Pager ☐ Office Email address: | |
| | | | Eman au | iii 035. |
| Occupational Position: | | | <u> </u> | |
| ☐ Faculty ☐ Physician ☐ Sta | ff Student Other: | | | |
| Project responsibilities: | | | | |
| Obtain consent from subjects | Provide access to patient pop | oulation 🗌 Oth | er: | |
| Conflict of Interest: | | | | |
| Does this person have a reportable | e conflict as defined in Section 1 | 1 of the applicat | tion? | |
| ∑ Yes ☐ No | | | | T |
| Required CITI Human Subjection | | | | HIPAA TRAINING |
| Date (Month/Year) CITI comp | pleted (either initial or refresh | er course): | | Check box below if HIPAA training is required. |
| 4/14 | | | | HIPAA Required – Data contains PHI |
| Note: The IRB requires researcher | | | | |
| Training | course. For more information on training requirements see IF | | | HIPAA Training completed through: |
| | | | | Other: |
| | Under: | | | |
| hutc0079 MD | | | | |
| Signature/Digital signature/x.500 | Signature/Digital signature/x.500 of Co-PI Title of Co-PI | | | |
| · | | | | |
| Research Staff | | | | |
| Research staff, including study coordinators, responsible for knowing and following the protocol, should be listed below. | | | | |
| Include any individual who will have responsibility for the consent process, direct data collection from subjects, or follow-up. | | | | |
| Study Staff Name (Last name, First name MI): Highest Earned Degree: | | | ed Degree: | |
| Cohen, Melissa | | | | |
| Affiliation and contact information | | | | |
| University of Minnesota (complete contact info section 1 Gillette (complete contact info section 2 only) | | | | |
| Fairview (complete contact | info section 2 only) | Other | (complete | contact info section 2 only) |
| Required Contact information | U of M Internet ID (x.500): cohen045 | | | |

| Section 1 - U of M only | U of M Employee/student ID Number: | | | |
|---|---|---|---|---|
| | University Department: | Anasthasialagy | | |
| | omversity Departments | nt: Anesthesiology | | |
| Required contact information | Address: Phon | | | e number: |
| Section 2 Non-U of M only | | | | |
| | | | ☐Mobile [ | ☐ Pager ☐Office |
| | | | Email addı | ress: |
| Occupational Position: | | | | |
| ☐ Faculty ☐ Physician ☐ Res | earch Coordinator Staff S | tudent 🔲 O | ther: | |
| Project responsibilities: | <del></del> | | | |
| Obtain consent from subjects | Other: | | | |
| Conflict of Interest: Does this per | son have a reportable conflict as | defined in Se | ction 11 of the | application? |
| ☐ Yes ⊠ No | | | | |
| Should This Person Be Copied | <u> </u> | es No | | |
| Required CITI Human Subje | | | | HIPAA TRAINING |
| Date (Month/Year) CITI comp | leted (either initial or refreshe | r course): | | Check box below if HIPAA training is required. |
| | | | _ | HIPAA Required – Data contains PHI |
| Note: The IRB requires researcher completion of initial course. For | | | | · |
| completion of mittal course. For | more imprination on training req | an ements set | <u>into Franing</u> | HIPAA Training completed through: MUMN |
| | | | | Other: |
| | | other. | | |
| Study Staff Name (Last name, Firs | st name MI): | | Highest Earne | d Degree: |
| Bryant-Huppert, Joe | | | MS | |
| Affiliation and contact inform | | | | |
| University of Minnesota (coonly) | omplete contact info section 1 | Gill | ette (complete | e contact info section 2 only) |
| Fairview (complete contact | info section 2 only) | Oth | er (complete c | contact info section 2 only) |
| Required Contact information | ntact information U of M Internet ID (x.500): hupp0037 | | | |
| Section 1 - U of M only | U of M Employee/student | t 2973892 | | |
| | ID Number: | | | |
| | University Department: | Anesthesiology, Medical student at Medical school | | |
| | 7cst.res.orogy, Medical stadelit at Medical School | | | |
| Required contact information | Address: | <u> </u> | Phone num | iber: |
| Section 2 Non-U of M only | | | | |
| | | | ☐Mobile [ | ☐ Pager ☐Office |
| | | | Email addı | ress: |

| Occupational Position: | |
|---|---|
| ☐ Faculty ☐ Physician ☐ Research Coordinator ☐ Staff ☒ Student ☐ Other: | |
| Project responsibilities: | |
| ☐ Obtain consent from subjects ☒ Other: asssist with data collection | |
| Conflict of Interest: Does this person have a reportable conflict as defined in Section 11 of the a | pplication? |
| ☐ Yes ☐ No | |
| Should This Person Be Copied on All Correspondence? Yes No | |
| Required CITI Human Subjects Training | HIPAA TRAINING |
| Date (Month/Year) CITI completed (either initial or refresher course): | Check box below if HIPAA training is |
| 07/15 required. | |
| Note: The IRB requires researchers to complete refreshers courses every three years after | HIPAA Required – Data contains PHI |
| completion of initial course. For more information on training requirements see IRB Training | HIPAA Training completed through: |
| | <b>⊠</b> UMN |
| | Other: |